CLINICAL TRIAL: NCT03335891
Title: The Effects of Core Stabilization Training on Dynamic Balance and Pulmonary Parameters Among Patients With Asthma: A Randomized Controlled Trial
Brief Title: The Effects of Core Stabilization Training Among Patients With Asthma: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif Develi, Teaching Assistant, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yeditepe University
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: asthma education program; balance; core stabilization exercises
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Asthma Education Program Breathing Exercises Core Stabilization Exercises
  Interventions: Procedure: Core Stabilization Exercises; Procedure: Control
- Control Group (Active Comparator): Asthma Education Program Breathing Exercises
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Core Stabilization Exercises — Volunteers received an asthma education program and trained for diaphragmatic, pursed lip breathing exercises as well as participated in the core stabilization exercises program.
  Arms: Training Group
Procedure: Control — Volunteers received an asthma education program and trained for diaphragmatic andpursed lip breathing exercises

SUMMARY:
Objective: To investigate the effectiveness of core stabilization exercises combined with the patient education program (AEP) and breathing exercises in patients with asthma.

Design: A randomized controlled study Setting: Chest diseases clinic of a university hospital. Subjects: The study sample consists of 26-68 years old asthma patients who were diagnosed at least 6 month prior to the study.

Interventions: All subjects were included in the asthma education program (AEP) and both groups were trained for diaphragmatic and pursed lip breathing exercises (2times/wk. 6-week duration at clinic). The core stabilization program was applied twice a week for a duration of 6 weeks in TG.

Main Measures: Spirometry, maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP), International Physical Activity Questionnaire Short Form (IPAQ), Hospital Anxiety and Depression Scale(HADS), Asthma Quality of Life Questionnaire(AQOL), Six-minute walking test(6MWT), Prokin PK200, Italy were used to evaluate feasibility of interventions.

DETAILED DESCRIPTION:
All volunteers received an asthma education program (AEP) and trained for diaphragmatic and pursed lip breathing exercises. Additionally, the TG participated in the core stabilization exercises program combined with AEP and breathing exercises. Data were collected from all the patients at baseline and post interventions (6 week) by the same physiotherapist who also supervised the exercise sessions.

All subjects were included in the asthma education program (AEP). AEP was performed at least once for approximately 20 minutes via face to face interviews. Education topics covered description of asthma, physiological changes of lungs, risk factors, treatment methods, relaxation positions to reduce dyspnea and usage of a specific inhaler. Breathing exercises were comprised of instructing breathing control, diaphragmatic breathing and pursed lip breathing exercises. Participants attended breathing exercises training for 2 days at the clinic under the supervision of a physiotherapist and 3 days at home as a home-exercise program. Total duration of breathing exercises lasted for 6 weeks. TG performed core stabilization exercises combined with breathing control for 2 days/a week for the duration of 6 weeks under the supervision of a physiotherapist at the clinic. Basic knowledges on spine, muscles of core stabilization and working principle of diaphragm and biofeedback unit (SPB) (Chattanooga Stabilizer Pressure Biofeedback, USA) were explained before the training. The SPB consists of an inflation pump and a cell like sphygmomanometer, which reflects body spinal movement in terms of mmHg by changing pressure in air filled cells. The SPB was placed under the lumbar 5th vertebra and patients attempted to maintain their core stability performing neutral zones at the settled level of 40 mmHg pressure. Furthermore, physiotherapist tried to improve thoracolumbar awareness by following changes from SPB and volunteers assured a constant lumbar position during upper and lower extremity movements combined with diaphragmatic movements. The 6 week exercise protocol emphasized core muscle co-contraction in hook-lying position with a flat cushion between two knees to provide integration between the pelvic floor muscles and diaphragm. Subsequently, exercises progressed as diaphragmatic breathing, flexion of both shoulder with breathing control and extending knees bilaterally with breathing control. Moreover, the hold time and the number of repetitions were increased from 5 repeats x 1 set to 5 repeats x 4 sets and each session lasted 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participating to the study in a voluntary basis.
* Being 18 years old and upper
* Getting diagnosed with asthma at least 6 months before.

Exclusion Criteria:

* Having an asthma attack in last 2 weeks.
* Having physical and/or mental disability.
* Having visual, hearing and/or verbal impairments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure | Six Weeks
  The Micro Medical Micro RPM, England respiratory pressure meter was used to measure respiratory muscle strength
Functional Capacity Test | Six Weeks
  The Six Minute Walking Test was used to evaluate functional capacity of volunteers. 6MWT was performed on a 30 meter corridor in the clinic according to American Thoracic Society guidelines. Walking distance was calculated.
Forced vital capacity in 1 second (FEV1) | Six Weeks
  Medical International Research Spirodoc® Spiro, Italy brand named spirometry was used to evaluate pulmonary functions of volunteers.
Quality of life | Six Weeks
  Asthma Quality of Life Scale (AQOL) was utilized to assess quality of life of participants over two weeks prior to the interview which was validated for the Turkish population.l
Maximum Expiratory Pressure | Six Weeks
  The Micro Medical Micro RPM, England respiratory pressure meter was used to measure respiratory muscle strength
Functional Vital Capacity (FVC) | Six Weeks
  Medical International Research Spirodoc® Spiro, Italy brand named spirometry was used to evaluate pulmonary functions of volunteers.
Tiffeneau Ratio (FEV1/FVC) | Six Weeks
  Medical International Research Spirodoc® Spiro, Italy brand named spirometry was used to evaluate pulmonary functions of volunteers.
Forced Expiratory Flow from 25 % to 75 % of Vital Capacity (FEF25-75) | Six Weeks
  Medical International Research Spirodoc® Spiro, Italy brand named spirometry was used to evaluate pulmonary functions of volunteers.

SECONDARY OUTCOMES:
Physical Activity | Six Weeks
  International Physical Activity Questionnaire Short Form (IPAQ) was used to determine physical activity status.The total score of IPAQ is calculated by summation of the duration (in minutes) and frequency (days) of three physical activities.
Depression level | Six Weeks
  The valid and reliable version of the Hospital Anxiety and Depression Scale (HADS) for the Turkish population was utilized to determine depression level.
Anxiety level | Six Weeks
  The valid and reliable version of the Hospital Anxiety and Depression Scale (HADS) for the Turkish population was utilized to determine anxiety level.
Dynamic balance | Six Weeks
  Dynamic balance alterations of the subjects were assessed by TechnoBody Prokin PK 200 (PK), Italy dynamic balance instrument. PK is a circular mobile balance assessment platform like conventional rocker board. PK transmits data from platform to the computer with a wireless transmitter and it can detect each single angular movement with a chip inside the platform. Additionally, PK has four different applicators (easy, medium, hard and rectangular) to place under the mobile platform. The bipedal position for 30 seconds with the easy applicator during the dynamic balance test was used. PK is connected to a computer; in this way each single movement is recorded by a computer in real time mode.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Develi, M.Sc., Principal Investigator — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Feryal Subasi, Professor, Study Chair — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Göksen Kuran Aslan, PhD, Study Chair — Istanbul University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Zuleyha Kaya Bingol, MD, Associate Professor, Study Director — Chest Medicine Outpatient Clinic of Istanbul University, Istanbul Medical Faculty

IPD SHARING:
Plan to Share IPD: No